CLINICAL TRIAL: NCT02376153
Title: Air Barrier System for the Prevention of Prosthesis-related Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nimbic Systems, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ABS004-H-35894
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Prosthesis-Related Infections
MeSH Terms: conditions — Prosthesis-Related Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABS deployed and active (Experimental): Air Barrier System (ABS) will be deployed onto the surgical field and activated.
  Interventions: Device: ABS deployed and active
- ABS deployed and NOT active (Sham Comparator): Air Barrier System (ABS) will be deployed onto the surgical field and NOT activated. This is a sham comparator to reduce the influence of the presence of the device and provide user blinding.
  Interventions: Device: ABS deployed and NOT active

INTERVENTIONS:
Device: ABS deployed and active — ABS is deployed onto surgical field and is turned on.
  Arms: ABS deployed and active
Device: ABS deployed and NOT active — ABS is deployed onto surgical field and is NOT turned on.
  Arms: ABS deployed and NOT active

SUMMARY:
This is a prospective, randomized, blinded clinical trial to determine if the Air Barrier System device reduces the incidence of surgical site infection after total hip replacement, acetabular repair, posterior spinal fusion, and prosthetic vascular graft procedures.

DETAILED DESCRIPTION:
This project is an evaluation of a novel device, the Air Barrier System (ABS), to reduce the risk of prosthesis-related surgical site infection in a multi-center clinical trial. The ABS shields surgical incisions intra-operatively by creating a field of high-purity air surrounding an incision that prevents airborne microorganisms from entering the incision.

This research will evaluate ABS performance in a prospective, randomized, blinded multi-center trial. The surgical procedures studied will include total hip arthroplasty, trauma-related acetabula reconstruction, posterior instrumented spine fusion, and prosthetic vascular graft procedures. Patients will be enrolled during the first two years of the study, and CDC guidelines require a one year follow-up period to monitor patients for potential prosthesis-related infections.

ELIGIBILITY:
Inclusion Criteria:

* Total hip arthroplasty;
* Acetabular repair with instrumentation;
* Posterior lumbar, cervical, or thoracic (up to and including 6 vertebral levels) spine fusion with instrumentation and vascular prosthetic graft implantation.

Exclusion Criteria:

* History of prior prosthesis infection;
* Active infection;
* Open traumatic wounds as is the case after some acetabular fractures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 816 (Estimated)
Dates: Start 2015-04-24 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Clinical incidence of surgical site infection | One-year post surgery
  Subjects are followed for one year post-surgery for onset of prosthesis-related infections .

CONTACTS AND LOCATIONS:
Overall Officials: Sean Self, Principal Investigator — Investigator
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan.